CLINICAL TRIAL: NCT05404685
Title: Randomised Study to Assess the Feasibility and Outcomes of Robotic Assisted Partial Nephrectomy in Low Pressure With AirSeal
Brief Title: Partial Nephrectomy in Low Pressure
Acronym: P-NeLoP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CHUBX 2020/62
Record Dates: First submitted 2022-04-27; First posted 2022-06-03 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Kidney Tumors Treated With Minimally Invasive Surgery
Keywords: kidney cancer; kidney tumor; robotic surgery; urology
MeSH Terms: conditions — Kidney Neoplasms; Carcinoma, Renal Cell

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: The randomization list is drawn up by the statistician of the Center for Methodology and Data Management (USMR of the Bordeaux University Hospital) before starting the research.
  The numbers of the 2 strategy groups are balanced with a 1:1 ratio. The randomization will be stratified on the study centers and a detailed description of the analgesia practices of each center will be made at the beginning of the study.
  The randomization will be done when the patient is under general anesthesia. Patients will not be told which group they have been randomized to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transperitoneal RAPN with AirSeal system set to 7mmH. (Experimental): Patient with Low Pressure Robotic Assisted Partial Nephrectomy at 7mm Hg
  Interventions: Device: Low insufflation pressure (7mm Hg) for Robotic Assisted Partial Nephrectomy
- transperitoneal RAPN with AirSeal system set to standard insufflation pressure (12mmHg) (Active Comparator): Control arm : Patient with standard insufflation pressure of 12 mm Hg
  Interventions: Device: Standard insufflation pressure (12mm Hg) for Robotic Assisted Partial Nephrectomy

INTERVENTIONS:
Device: Low insufflation pressure (7mm Hg) for Robotic Assisted Partial Nephrectomy — Use of insufflation pressure at 7 mm Hg. The groups will differ only with respect to the insufflation pressure level set on the AirSeal® system.
  The level of pressure will be adjusted at the beginning of the surgery, after placement of the trocars, in accordance with the result of the randomization.
  Arms: Transperitoneal RAPN with AirSeal system set to 7mmH.
Device: Standard insufflation pressure (12mm Hg) for Robotic Assisted Partial Nephrectomy — Use of insufflation pressure at 12 mm Hg. The groups will differ only with respect to the insufflation pressure level set on the AirSeal® system.
  The level of pressure will be adjusted at the beginning of the surgery, after placement of the trocars, in accordance with the result of the randomization.
  Arms: transperitoneal RAPN with AirSeal system set to standard insufflation pressure (12mmHg)

SUMMARY:
The main objective is to prospectively assess the impact of low insufflation pressure using AirSeal system (7mm Hg) during RAPN on post-operative patient pain (main location and intensity), 24 hours after surgery. The study will be conducted among 15 centers of the French research network on kidney cancer UroCCR.

DETAILED DESCRIPTION:
Minimally invasive route for PN is recommended to offer patients ERAS and day-case pathways leading to the best possible recovery. In this setting, pain management is crucial and every innovation supposed to offer a benefit has to be assessed. For transperitoneal laparoscopic procedures, the level and stability of the insufflation pressure will influence the quality of the pneumoperitoneum and may impact the feasibility of the surgery as well as intra and post-operative outcomes. It is universally recognized that the lower insufflation pressure, the better. However, a balance has usually to be found between technical feasibility of the surgery and lowest acceptable insufflation pressure. The AirSeal system aims to generate a stable pneumoperitoneum even in case of active gaz succion by the surgeon's assistant. The investigators then hypothesize that RAPN would be feasible and safe even in low pressure (7mm Hg) and may decrease post-operative patients' pain.

The investigators plan to describe the feasibility of Low Pressure RAPN at 7mm Hg (LP-RAPN) and assess its intra and post-operative outcomes including pain and recovery on a patient perspective. This will be achieved comparatively to RAPN performed at standard insufflation pressure of 12 mm Hg and through a single blinded randomized trial design.

The project has been developed and will be conducted within the framework of the French research network on kidney cancer UroCCR (www.uroccr.fr). INCa has been supporting this multidisciplinary network since 2011 and the web-based shared clinical and biological national database on kidney cancer UroCCR will be used.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female aged of 18 and over
* Planned transperitoneal RAPN for tumor with AirSeal system.
* Affiliation to or beneficiary of the French social security
* Patient in capacity and willing to accurately report pain-killer intakes in the first postoperative 7 days.
* Free, informed and written consent signed by the patient and the investigating physician (at the latest on the day of inclusion and before any examination required by the research).

Exclusion criteria:

* Daily chronic pain-killers intake for another indication than the kidney tumor and intended to be maintained at the time of surgery
* Person deprived of liberty
* Person under trusteeship, curatorship or legal guardianship
* Refusal of consent or participation in the UroCCR project and the P-NeLoP ancillary trial

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Actual)
Dates: Start 2022-10-04 (Actual); Primary Completion 2024-04-29 (Actual); Study Completion 2024-04-29 (Actual)

PRIMARY OUTCOMES:
Intensity of post-operative pain | 24 hours after surgery
  intensity of pain measured by a numeric analogic scale (between 0 and 10)

SECONDARY OUTCOMES:
Number of clamp procedures. | at surgery
  Determination of the number of off-clamp procedures and the number of on-clamp procedures (type and length of clamping)
Main location and intensity of post-operative pain. | 6 hours and 48 hours after surgery
  Determination of main location and intensity (visual analogic scale) of post operative pain (minimum=0 correspond to worse outcome; maximum =10 correspond to better outcome)
Length of surgery | up to 30 Days
  determination of length of surgery in minutes
Estimated blood loss and intra-operative transfusion | at surgery
  Estimated blood loss (mL) and intra-operative transfusion

OTHER OUTCOMES:
Plateau Pressure and PETCO2 60 minutes after incision | at surgery
Length of Hospital stay (days) | up to 30 days after surgery
  Determination of Length of Hospital stay (days)
Number and Clavien-Dindo classification of intra and post-operative complications up to 30 days after surgery | up to 30 days after surgery
Pain-killer intake scoring during the first post-operative week (7days) | up to 7 days after surgery
Minutes between end of surgery and first time out of bed | up to Day 2
Minutes between end of surgery and resumption of feeding | up to Day 2 after surgery
Minutes between end of surgery and resumption of bowel function (stools) | up to day 7 after surgery
Cost difference between the two arms (€) | at surgery
Minutes between end of surgery and resumption of bowel function (gaz) | up to day 2 after surgery

CONTACTS AND LOCATIONS:
Locations (15):
- France (15):
  - CHU d'Angers, Angers
  - Centre Hospitalier Universitaire de Bordeaux, Bordeaux
  - CHU de Caen, Caen
  - Hopital Henri-Mondor, Créteil
  - Hôpital Claude Huriez, Lille
  - Institut Paoli-Calmettes, Marseille
  - CHU de Nice, Nice
  - Hôpital Pitié-Salpétrière, Paris
  - Hôpital bicêtre, Paris
  - Polyclinique Francheville Périgueux, Périgueux
  - CHU de Poitiers, Poitiers
  - Clinique La Croix du Sud, Quint-Fonsegrives
  - CHU de Rennes, Rennes
  - CHRU de Strasbourg, Strasbourg
  - CHU de Tours, Tours

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Margue G, Bigot P, Ingels A, Roupret M, Waeckel T, Long JA, Pignot G, Bensalah K, Lang H, Olivier J, Bruyere F, Durand M, Beauval JB, Mallet R, Parier B, De La Taille A, Bernhard JC. Clinical trial protocol for P-NeLoP: a randomized controlled trial comparing the feasibility and outcomes of robot-assisted partial nephrectomy with low insufflation pressure using AirSeal versus standard insufflation pressure (UroCCR no. 85 study). Trials. 2023 Aug 19;24(1):545. doi: 10.1186/s13063-023-07533-4. PMID 37596613